CLINICAL TRIAL: NCT07187362
Title: Comparison of Posterior Cellular Bonegraft Options for Single Level Lumbar Spinal Fusion: A Randomized Trial
Brief Title: Comparison of Posterior Cellular Bonegraft Options for Single Level Lumbar Spinal Fusion
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Midwest Spine & Brain Institute (Other)
Responsible Party: Principal Investigator, Glenn Buttermann, MS, MD, Medical Doctor, Principle Investigator, Midwest Spine & Brain Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HE 15 10 002
Record Dates: First submitted 2025-09-18; First posted 2025-09-23 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Disc Degenerative Disease; Spine Fusion for Degenerative Spine Disease
Keywords: surgery; allograft bone
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Intervention Model Description: randomized, prospective
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- iliac bone graft (Active Comparator): old standard of care
  Interventions: Biological: Use iliac bone graft
- Bone morphogenetic protein (Experimental): Known osteoinductive bone graph
  Interventions: Biological: use bone morphogenetic protein
- MSCs from bone allograft (Experimental): extracted MSCs from human cadeveric bone
  Interventions: Biological: use bone derived allograft MSCs
- MSCs from amnion/placental tissue (Experimental): MSCs derived from human afterbirth tissue
  Interventions: Biological: Use amnion/placental derived MSCs
- MSCs from human adipose tissue (Experimental): MSCs derived from human fat
  Interventions: Biological: Use adipose tissue derived MSCs

INTERVENTIONS:
Biological: Use iliac bone graft
  Arms: iliac bone graft
Biological: use bone morphogenetic protein
  Arms: Bone morphogenetic protein
Biological: use bone derived allograft MSCs
  Arms: MSCs from bone allograft
Biological: Use adipose tissue derived MSCs
  Arms: MSCs from human adipose tissue
Biological: Use amnion/placental derived MSCs
  Arms: MSCs from amnion/placental tissue

SUMMARY:
This study involves the assessment of alternatives to iliac bone graft during spinal fusion surgery. Four types of bone graft alternatives are being compared to iliac bone graft during the posterior portion of an anterior/posterior one-level lumbar spinal fusion. If you choose to participate in this study, you will be randomized (like a flip of a coin) to receive either your own iliac bone graft, bone morphogenetic protein (BMP, made from proteins found in the human body that stimulate bone growth), or one of the following stem-cell based bone graft alternatives for the posterior portion of your fusion surgery:

* Orthofix Trinity-made from donor bone and bone marrow stem cells
* Allosource Allostem-made from donor bone and fat stem cells
* Nutech Nucel-made from donor bone and placenta (after birth) stem cells

Each bone graft alternatives has been approved by the United States Food and Drug Administration (FDA) and is commercially available with the exception that BMP application is considered "off-label". That is, BMP it is not approved for this indication, it is currently indicated for anterior fusion. The volume of bone graft that you will receive is the same for each graph type (approximately 5cc). Approximately 150 patients from the Midwest Spine and Brain Institute are expected to be enrolled in this study. If you choose to take part, your participation will last about 2+ year.

At approximately 9 - 15 months after your surgery, you will be asked to return to the Midwest Spine and Brain Institute to undergo a limited CT scan of the fusion level to determine how you are healing. Your pain level and functional ability will also be evaluated at this visit.

DETAILED DESCRIPTION:
Consecutive patients who are surgical candidates for a one-level anterior/posterior lumbar fusion are eligible for inclusion into the study. Inclusion criteria included:

* 18 to 65 years of age.
* Primary degenerative disc disease of one level with or without prior decompression.
* None or up to moderate stenosis that could be treated with a laminotomy
* degenerative spondylolisthesis grade 2 or less.

Exclusion criteria:

* More than single level symptomatic degenerative disc disease.
* Advanced stenosis that needed extensive laminectomy for adequate decompression.
* Lytic spondylolisthesis.

The study proposal underwent IRB review (HealthEast IRB #1510002). All the participants provided written informed consent. After completing IRB approved consent, patients were randomized, by computer generated program, to 5cc IBG or one of 5 other types of PSF osteoinductive bone graft alternatives: bone morphogenic protein (BMP, small Infuse, Medtronic, Memphis, TN), autologous concentrated bone marrow aspirate (BMA) from the iliac crest (combined with 5cc Allo chips), allograft bone marrow derived stem cells (cAlloBone, 5.3cc Trinity Elite, Orthofix, Lewisville, TX), fat derived allograft stem cells (Allostem, AlloSource, Centennial, CO) combined with 5cc morcelized cancellous allograft (cAlloFat), or placental derived allograft stem cells (NuCel, Nutech, Birmingham, Alabama) combined with 5cc morcelized cancellous allograft (cAlloAm). A historical control group of 5cc cancellous freeze-dried allograft (Allo) was used as an inert "negative" control group. There are 27 patients in each group. All anterior fusions used BMP (small Infuse). The decortication technique of the posterior fusion is identical for all patients. All patients have identical fixation instrumentation implanted (anterior lumbar plate and posterior facet screws). Posterior fusions were instrumented to eliminate posterior micromotion and subsequent pseudarthrosis as a confounding variable. All the fusion procedures were performed by the lead author to ensure a uniform surgical technique across all bone graft type groups. Therefore, the surgical technique is as uniform as practically possible to minimize confounding variables related to the surgery with the only variable being the various posterior fusion bone graft materials. Patients are blinded to the posterior type of bone graft. The volume of bone graft is the same for each type, approximately 5cc.

Postoperatively, all patients are followed for a minimum of 2 years. During this time radiographs and lumbar Thin-cut CT scans of the fused level are obtained at approximately one year postoperatively to assess fusion success of both anterior and posterior spinal columns. Specifically for the posterior fusion, if only a unilateral fusion was identified, the fusion was tallied as half fused. The limited (to the levels fused) CT scan had 2.88 mSv radiation exposure, or similar to one year's worth of background radiation. Radiographs at >2 years are reviewed for progressive loss of adjacent segment disc height for assessment of adjacent level degeneration. Secondary endpoints of clinical outcomes are assessed pre- and postoperatively with multiple outcome instruments: visual analog scales (VAS, 0 to 10 scale with greater value is worse pain) for back and leg pain; pain drawing; Oswestry disability index (ODI, 0 to 100 scale with greater value is worse disability); pain medication usage (non-opioid and opioids); and patient self-assessment of procedure success over a minimum 2-year follow-up period. Outcome results are entered by office personnel (blinded to the type of bone graft) into computer spreadsheets, with the treating surgeon blinded to these results. The historical control group consisted of retrospective cohort of consecutive patients which fit the inclusion/exclusion criteria and had their PSF with freeze-dried allograft morcelized bone. Additional surgeries were tracked for all groups, including pseudarthrosis repair, adjacent level decompression, adjacent-level fusion extension, spinal cord stimulator implantation, and posterior instrumentation removal.

ELIGIBILITY:
Inclusion Criteria: Single level lumbar degenerative disc disease -

Exclusion Criteria: Degenerative spondylolisthesis >grade 1, lytic spondyolisthesis, infection, stenosis requiring laminectomy, cancer, scoliosis, pregnancy

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2015-10-13 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Solid spinal fusion | 1 year
  Assessed by thin cut CT scan

SECONDARY OUTCOMES:
Pain and disability | 1, 2 and 2+ years
  Self-assessment questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Glenn R BUTTERMANN, Principal Investigator — Midwest Spine & Brain Institute

IPD SHARING:
Plan to Share IPD: No
Trial start date began prior to 2017

DOCUMENTS (2):
  • Study Protocol (2015-10-03): https://cdn.clinicaltrials.gov/large-docs/62/NCT07187362/Prot_000.pdf
  • Informed Consent Form (2015-10-12): https://cdn.clinicaltrials.gov/large-docs/62/NCT07187362/ICF_001.pdf